CLINICAL TRIAL: NCT03701230
Title: Safety and Efficacy of Low Temperature Rota-flush Solution for the Treatment of RA-related Myocardial Injury in Patients With Severe Calcified Lesion Undergoing Rotational Atherectomy (RA) (LOTA-II)
Brief Title: Safety and Efficacy of Low Temperature Rota-flush Solution in Patients With Severe Calcified Lesion (LOTA-II)
Acronym: LOTA-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20180713-04
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Injury
Keywords: low temperature; rota-flush solution; RA-related myocardial injury; severe calcified lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low temperature rota-flush solution (Experimental): A total of 66 patients are assigned to low temperature rota-flush solution group after randomization schedule.
  Interventions: Other: low temperature rota-flush solution
- room temperature rota-flush solution (No Intervention): A total of 66 patients are assigned to room temperature rota-flush solution group after randomization schedule.

INTERVENTIONS:
Other: low temperature rota-flush solution — Patients with severe calcified lesions undergoing RA were performed with low temperature rota-flush solution. The investigators used thermal insulation equipment to keep rota-flush solution at 0～5℃. The EKG and blood pressure were monitored during the RA procedure. After RA, the investigators monitored levels of myocardial injury biomarkers for 3 days every 8 hours.
  Arms: low temperature rota-flush solution

SUMMARY:
Calcified lesions related to coronary artery are a type of atherosclerosis, accompanied by severe calcified lesions of the stenosis, which is a difficult point for PCI interventional therapy. Calcified lesions have poor response to balloon dilatation and the device can not be successfully placed, which reduce the success rate of operation. Furthermore, the stent is under-expanded and the adherence is poor, which significantly increases the incidence of major adverse cardiovascular events (MACEs).

Intracoronary rotational atherectomy (RA) was developed by David Auth in the early 1980s. In 1988, Bertrand has completed the first case of coronary RA. RA was recommended for treatment of severe calcified lesions in ACC/AHA Guidelines for Coronary Interventional Therapy in 2011 (IIa, C). However, many studies have found that the incidence of RA-related myocardial injury is relatively high, and affect the efficacy of RA and prognosis in patients with severe calcified lesions. It has been reported that 58 consecutive patients with stable angina requiring PCI with RA to a calcified coronary lesion have 68% 5-fold increase in high sensitivity troponin after RA. The objective of this randomized control trial is to gain a clinical insight on the use of low temperature rota-flush solution for the treatment of RA-related myocardial injury in patients with heavy calcified lesions. The primary objective is assess efficacy and safety of low temperature rota-flush solution for the treatment of RA-related myocardial injury in patients with severe calcified lesions.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, randomized and prospective study aiming to compare the incidence rate of RA-related myocardial injury indicated by change in levels of myocardial injury biomarkers (such as TNI and CK-MB) between low temperature rota-flush solution group and room temperature rota-flush solution group. Based on previous study, the incidence rate of RA-related myocardial injury is 68.0 % in patients with severe calcified lesions undergoing PCI. And in our study the expected incidence rate of RA-related myocardial injury is up to 34.0 % in patients with severe calcified lesions undergoing PCI after treatment with low temperature rota-flush solution. Moreover, the investigators estimated 10% loss follow-up of these patients in each arm. As a result, a total of 132 patients with heavy calcified lesions were required, and with 66 patients per group as a ratio of 1:1 randomization.

ELIGIBILITY:
Inclusion Criteria:

* De novo lesions
* Severe coronary calcified lesion (detected by CAG, IVUS or OCT)
* New generation drug eluting stent implantation
* Only single coronary artery treated at this time

Exclusion Criteria:

* Those who meet the diagnostic criteria of acute myocardial infarction
* Patients with cardio-genic shock
* Patients with multiple organ failure
* Patients allergic to contrast
* Patients who can not tolerate dual antiplatelet therapy
* Patients who can't tolerate anticoagulation
* Recently infected patients
* Patients with hepatorenal dysfunction
* Thrombotic lesion of coronary artery
* Spontaneous coronary dissection
* Patients with drug coated balloon treatment
* Patients with bioabsorbable vascular scaffold implantation
* Previous percutaneous coronary intervention or coronary artery bypass graft
* Patients with active stage of autoimmune disease
* Patients with complex coronary bifurcation requiring two stent strategy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
the incidence rate of RA-related myocardial injury in patients with severe calcified lesions 3 days after RA. | 3 days after RA
  the incidence rate of RA-related myocardial injury indicated by the changes in myocardial injury biomarkers (such as TNI and CK-MB) between low temperature rota-flush solution and room temperature rota-flush solution groups in patients with severe calcified lesions 3 days after RA.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ye, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (8):
- China (8):
  - The Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First People's Hospital of Chuzhou, Chuzhou, Anhui
  - MingGuang People's Hospital, Chuzhou, Anhui
  - The Second People's Hospital of Huaian, Huaian, Jiangsu
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The People's hospital of Yixing, Yixing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mosseri M, Satler LF, Pichard AD, Waksman R. Impact of vessel calcification on outcomes after coronary stenting. Cardiovasc Revasc Med. 2005 Oct-Dec;6(4):147-53. doi: 10.1016/j.carrev.2005.08.008. PMID 16326375
- [Background] Shan P, Mintz GS, Witzenbichler B, Metzger DC, Rinaldi MJ, Duffy PL, Weisz G, Stuckey TD, Brodie BR, Genereux P, Crowley A, Kirtane AJ, Stone GW, Maehara A. Does calcium burden impact culprit lesion morphology and clinical results? An ADAPT-DES IVUS substudy. Int J Cardiol. 2017 Dec 1;248:97-102. doi: 10.1016/j.ijcard.2017.08.028. Epub 2017 Aug 12. PMID 28818353
- [Background] McEntegart M, Corcoran D, Carrick D, Clerfond G, Sidik N, Collison D, Robertson KR, Shaukat A, Watkins S, Rocchicholi PR, Eteiba H, Petrie MP, Lindsay MM, Oldroyd KG, Berry C. Incidence of procedural myocardial infarction and cardiac magnetic resonance imaging-detected myocardial injury following percutaneous coronary intervention with rotational atherectomy. EuroIntervention. 2018 Sep 20;14(7):819-823. doi: 10.4244/EIJ-D-17-01077. No abstract available. PMID 29741483
- [Derived] You W, Wu XQ, Wu ZM, Wang YF, Shen TT, Tang B, Xu T, Ying LH, Pan DF, Yang S, Yin DL, Ye F. Safety and efficacy of low-temperature RA-flush solution in patients with moderate-to-severe calcified lesions (LOTA-II): a randomized, double-blind, multicenter study. Sci Rep. 2025 May 25;15(1):18280. doi: 10.1038/s41598-025-02799-x. PMID 40415011